CLINICAL TRIAL: NCT04286945
Title: Lateral Rectus Muscle Tendon Elongation by an Auto Graft From the Resected Medial Rectus Muscle as a Monocular Surgery for Large Angle Sensory Exotropia
Brief Title: Lateral Rectus Muscle Tendon Elongation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Heba Shafik, Principal investigator, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21423
Record Dates: First submitted 2020-02-19; First posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Surgical Procedure, Unspecified; Ocular Discomfort; Strabismus, Divergent
Keywords: SENSORY EXOTROPIA; LATERAL RECTUS ELONGATION; AUTOGRAFT
MeSH Terms: conditions — Exotropia

STUDY DESIGN:
Intervention Model Description: PROSPECTIVE STUDY
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SENSORY EXOTROPIA PATIENTS WITH LARGE ANGLES . (Other): Patients with monocular low vision or loss of vision due to congenital or acquired cause with exodeviation of the poorly seeing eye ≥ 50PD, were included in the study.
  Interventions: Procedure: LATERAL RECTUS MUSCLE AUGMENTED RECESSION BY ELONGATION OF THE TENDON WITH AUTOGRAFT FROM RESECTED MEDIAL RECTUS MUSCLE

INTERVENTIONS:
Procedure: LATERAL RECTUS MUSCLE AUGMENTED RECESSION BY ELONGATION OF THE TENDON WITH AUTOGRAFT FROM RESECTED MEDIAL RECTUS MUSCLE — After resection of the medial rectus muscle, the resected segment is sutured to the lateral rectus muscle after dissection and marking to elongate and slaken the muscle then the elongated muscle is sutured to the sclera at the desired amount of conventional recession.
  Other Names: Lateral rectus elongation

SUMMARY:
To evaluate a technique using resected medial rectus muscle transplantation for elongation of Lateral rectus tendon as a monocular surgery for large angle sensory exotropia.

DETAILED DESCRIPTION:
A prospective study done in Tanta university in the period between January 2017 and June 2018.It included 16 patients with sensory exotropia ≥50PD. Full history was taken. Visual acuity, cycloplegic refraction and fundus exam of both eyes was performed prior to surgery. Strabismus angles were measured at near and distance by alternate prism cover test. Any limitation of adduction or abduction was scaled from -4 to 0. Patients were followed for 6 months.

SURGICAL PROCEDURE:

The MR muscle was dissected through a limbal incision. Two single arm 6-0 Vicryl sutures were placed at desired distance from the insertion as the routine resection of rectus muscle and another pair of 6-0 Vicryl was placed at the insertion. The muscle was then incised from its insertion, and the posteriorly (distally) placed 6-0 Vicryl sutures were passed through the original insertion. The resected segment is then put in saline. A vicryl 6-0 suture was tied at the LR muscle insertion. The muscle was incised from its insertion. Next, the stump of the resected segment was then sutured to the sclera at the desired position measured by the strabismus caliber according to the surgical dosage sufficient to correct the premeasured distant angle (taking into consideration the length of the added segment, which will be added to the amount of recession), and the distal end of this stump was sutured with the proximal end of LR with the 6-0 Vicryl already placed on the LR. Now the elongated muscle was sutured at desired site from the original insertion of LR as done in routine rectus muscle recession.

The patients were followed at 1day after surgery, 2 weeks, 3 month, and 6 months.

In each visit the distant angle of deviation was measured by prism cover test, any limitation of adduction and abduction was scaled, and patient satisfaction with results at last follow up was obtained, all results were recorded and tabulated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with monocular low vision or loss of vision due to congenital or acquired cause with exodeviation of the poorly seeing eye ≥ 50PD.

Exclusion Criteria:

* Patients with exotropia other than sensory type (alternating exotropia, intermittent exotropia)
* Angle of deviation less than 50 PD.
* visual acuity more than 0.2 decimal in affected eye .
* A or V pattern exotropia.
* Nystagmus .
* Refusal of surgery by the adult patients or caregiver of children.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Distant angle of deviation after surgical correction | 6month
  Measured by alternate prism cover test for near and far,which is considered successful if within10 prism diopter esotropia or exotropia.
limitation of adduction and abduction | 6month
  measured by a scale from -4 to 0; with-4 implying no adduction or abduction beyond midline, -3 implying for 75% deficit,-2 for 50% deficit,-1 for 25% deficit and 0 for full ductions.
patient satisfaction with the procedure | after 6 month
  score assesed by questionnaire of 3questions based on satisfaction with degree of alignment, aesthetic appearance, limitation of adduction and abduction. 0: I am not satisfied, 1: I am moderately satisfied, 2: I am satisfied, 3: I am very satisfied, and Iwould recommend it to another.
  Based on the score (0-3 unsatisfied, 4-6 moderately satisfied, 7-9 very satisfied).

IPD SHARING:
Plan to Share IPD: Yes
share data after publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: within 6 month of completion of the study
Access Criteria: after publication in a subspecialized journal reviewed by panel reviewers that has an open access on line

REFERENCES:
- [Derived] Shafik HM, Eldesouky MA, Elbakary MA, Elbedewy HA. Unilateral surgery for pediatric sensory exotropia: clinical characteristics and surgical results. BMC Ophthalmol. 2022 Dec 22;22(1):507. doi: 10.1186/s12886-022-02722-2. PMID 36550417